CLINICAL TRIAL: NCT00745511
Title: A Randomized, Multi-Center, Double Blind, 3 Arm, Phase I/II Pilot Study to Evaluate the Safety and Efficacy of Treatment With ORA102 Combined With Avastin (Bevacizumab) Versus Avastin Alone, in Patients With Neovascular Age Related Macular Degeneration (AMD)
Brief Title: Pilot Study to Evaluate the Safety and Efficacy of Treatment With ORA102 Combined With Avastin (Bevacizumab) Versus Avastin Alone, in Patients With Neovascular Age Related Macular Degeneration (AMD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ora Bio Ltd. (Industry)
Responsible Party: Yossi israeli, Ora Bio Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OB-DAMD-01
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Macular Degeneration
Keywords: AMD; Avastin; ORA102; macular degeneration; neo-vascular age related macular degeneration (AMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator)
  Interventions: Drug: ORA102 and Avastin
- 2 (Active Comparator)
  Interventions: Drug: ORA102 and Avastin
- 3 (Placebo Comparator)
  Interventions: Drug: Avastin

INTERVENTIONS:
Drug: ORA102 and Avastin — treatment with intravitreal injections of Avastin 1.25mg (0.05ml)and ORA102
  Arms: 1; 2
Drug: Avastin — treatment with intravitreal injections of Avastin 1.25mg (0.05ml)
  Arms: 3

SUMMARY:
This is s randomized, multi-center, double blind, 3 arm, phase I/II pilot study to evaluate the safety and efficacy of treatment with ORA102 combined with Avastin (Bevacizumab) versus Avastin alone, in patients with neo-vascular age related macular degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have provided informed consent, including signing of the informed consent form
* Subject who are able and willing to comply with the study protocol
* Subject must have best corrected visual acuity ETDRS between 20/40 to 20/320 in the study eye
* Subjects whose CNV lesion in the study eye contains more than 25% scarring and/or atrophy
* Women must be post-menopausal 1 year or surgically sterilized. If not, negative serum pregnancy test required within 14 days of randomization

Exclusion Criteria:

* Pregnant or lactating women
* Patients with severe myocardial disease or coronary occlusion
* Patients with severe personality disorder, suicidal risk or psychosis
* Patients with previous history of CVA
* Evidence for liver dysfunction - bilirubin level more than twice than upper limit of the normal value OR ALT/AST>1.5x upper limit of normal value
* Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contra-indicates the use of the investigational drugs or puts the patients in high risk for treatment related complications

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of ocular adverse events, including retinal detachment, increase in IOP, cataract, tearing of the retina, decrease in vision, RPE atrophy, and vitreous hemorrhage, will be evaluated. | 32 weeks

SECONDARY OUTCOMES:
Central Retinal thickness and presence of intra/sub-retinal fluid observed by OCT at week 32 | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Itay Chovers, MD, Principal Investigator — Hadassah Medical Organization
Locations (5):
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Carmel Medical Center, Haifa
  - Hadassah Medical center Israel, Jerusalem
  - Ziv Medical Center, Safed
  - Tel-Aviv Sourasky Medical Center, Tel Aviv